CLINICAL TRIAL: NCT04436367
Title: Retrospective Study of Patients With Severe Aplastic Anemia Who Developed High Risk Clonal Evolution With Chromosome 7 Abnormalities After Immunosuppressive Therapy
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920118; 20-H-N118
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Severe Aplastic Anemia
Keywords: Cytogenic Abnormality; Natural History
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- SAA patients with Monosomy 7: Severe Aplastic Anemia Patients who Developed High Risk Clonal Evolution with Chromosome 7 Abnormalities after Immunosuppressive Therapy

SUMMARY:
Background:

Severe aplastic anemia (SAA) is a form of bone marrow failure. It usually results from a

cytotoxic T cell attack on the marrow stem cell. Two treatments can be used for SAA. One is allogeneic hematopoietic stem cell transplant (HSCT). The other is immunosuppressive treatment (IST). In most cases, HSCT or IST works. But for some people, clonal evolution occurs after IST. One of the most common forms of clonal evolution is chromosome 7 abnormalities. These have a poor prognosis. HSCT can be used to treat them. Researchers do not know why clonal evolution happens. They want to look at data from past studies to learn more.

Objective:

To compare the data of people with SAA who developed chromosome 7 abnormalities between those who ultimately received HSCT versus those who received chemotherapy alone or supportive care.

Eligibility:

Adults and children with SAA who were enrolled on NHLBI protocol 12-H-0150, 06-H-0034, 03-H-0249, 03-H-0193, 00-H-0032, or 90-H-0146

Design:

This study uses data from past studies. The participants in those studies have allowed their data to be used in future research.

Researchers will review participants medical records. They will collect clinical data, such as notes, test results, and imaging scans. They will also collect the research data gathered as part of the original study.

Researchers will enter the data into an in-house database. It is password protected. All data will be kept in secure network drives or in sites that comply with NIH security rules.

Other studies may be added in the future.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a form of bone marrow failure in most cases is the result of a cytotoxic T cell attack on the marrow stem cell. It is effectively treated in most patients with either immunosuppressive treatment (IST) or allogeneic hematopoietic stem cell transplant (HSCT). However, after IST, 'clonal evolution' is a significant complication in about 15% of patients, presenting as either a new cytogenetic abnormality or morphological evidence of myeloid malignancy. In particular, the development of chromosome 7 abnormalities is considered high risk and is associated with poor prognosis. The optimal treatment of chromosome 7 abnormalities following SAA is not defined though HSCT is widely offered.

ELIGIBILITY:
* Subjects will not be recruited for this study. This is a retrospective chart review.

Patients who opted out of future use of data on their prior studies will be excluded from this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SAA Subjects who developed chromosome 7 abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Characteristics and outcomes of SAA patients who developed chromosome 7 abnormalities | Between the Period of 1990 to 2020
  To compare characteristics and outcomes of SAA patients who developed chromosome 7 abnormalities between those who ultimately received HSCT versus those who received chemotherapy alone or supportive care

SECONDARY OUTCOMES:
Clinical predictors for the development of chromosome 7 abnormalities such as age, gender, baseline laboratory value | Between the Period of 1990 to 2020
  To identify clinical predictors for the development of chromosome 7 abnormalities such as age, gender, baseline laboratory values, time from diagnosis to initial treatment, relapse, and number of IST treatments
Ascertain the natural history of patients with a chromosome 7 abnormality on karyotype | Between the Period of 1990 to 2020
  Ascertain the natural history of patients with a chromosome 7 abnormality on karyotype who were surveilled until the development of an overt myeloid neoplasm
Morphological predictors in the bone marrow for progression to an overt myeloid neoplasm | Between the Period of 1990 to 2020
  To identify morphological predictors in the bone marrow for progression to an overt myeloid neoplasm in those with without an overt myeloid neoplasm at the time of development of chromosome 7 abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Groarke, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States